CLINICAL TRIAL: NCT01687517
Title: Determination of the Efficacy and Safety of the Seasonal Influenza Vaccine Among Patients Suffering From Sarcoidosis.
Brief Title: Efficacy and Safety of Influenza Vaccine During Sarcoidosis
Acronym: SARCOVAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P110115
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Sarcoidosis; Influenza Vaccine
Keywords: sarcoidosis; healthy volunteers
MeSH Terms: conditions — Sarcoidosis; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient (Experimental): 90 patients suffering from sarcoidosis
  Interventions: Drug: Seasonal influenza vaccine available for the 2012-2013 vaccine campaign
- Volunteer (Active Comparator): 100 volunteers
  Interventions: Drug: Seasonal influenza vaccine available for the 2012-2013 vaccine campaign

INTERVENTIONS:
Drug: Seasonal influenza vaccine available for the 2012-2013 vaccine campaign — Single injection of the vaccine at D0 (0.5mL intra-muscularly or subcutaneous for patient under anticoagulant treatment)

SUMMARY:
Sarcoidosis is an inflammatory disease of unknown origin that can affect all organs, especially the lungs and mediastinum. Some location of sarcoidosis may require treatment with corticosteroids or immunosuppressors.Although seasonal influenza vaccination can be recommended in sarcoidosis in some subgroups at risk (respiratory failure, pulmonary fibrosis, age over 65, use of immunosuppressive therapy, etc ...), the investigators presently have no data on the efficacy and safety (absence of adverse reactions) of seasonal influenza vaccination in sarcoidosis.Especially it is not known whether the seasonal influenza vaccine provides the same rate and same type of vaccine response in sarcoidosis patients than in the general population. Similarly, it is unclear whether the vaccine response is modified by the severity of the disease and treatment with corticosteroids and immunosuppressors.Based on what is known in systemic lupus and rheumatoid arthritis, which are both inflammatory and autoimmune diseases, the investigators expect at best a 50% vaccine response in patients with sarcoidosis and a 85% vaccination response in healthy controls. The demonstration of a vaccine response could allow reconsidering new vaccine approaches in sarcoidosis.

DETAILED DESCRIPTION:
Data on vaccination in sarcoidosis are largely insufficient. It is thus unclear whether the vaccine response is modified according to the clinical phenotype of the disease and/or treatment with corticosteroids and immunosuppressants. However, sarcoidosis is accompanied by numerous disturbances of the immune system, including a tendency to anergy which may affect the efficacy of the vaccine, especially when the disease is active and severe. In addition, the tolerance of influenza vaccination in patients with sarcoidosis has not been studied yet.The influenza vaccination in sarcoidosis is a common practice among medical specialists who care for patients with sarcoidosis, either internists or lung specialists.. However, the practice of this vaccination is not based on scientific evidence, because there are no data establishing the efficacy and safety of influenza vaccination in sarcoidosis.Thus, it is possible that the influenza vaccine is less immunogenic in patients with sarcoidosis than in healthy adults, which may reduce the clinical effectiveness of vaccination. It therefore seems essential to determine the efficacy and safety of this vaccine, which is widely practiced. Poor efficiency could lead to the development of different vaccination strategies, based in particular on the administration of adjuvanted vaccines.

ELIGIBILITY:
Inclusion Criteria for patients:

* Age ≥ 18 and ≤ 65;
* Signature of informed consent
* Follow-up : six months following the influenza vaccination at D0
* Sarcoidosis diagnosed and histologically proven since at least 6 months
* unchanged treatment of Sarcoidosis for at least 3 months, except for the case of a decrease in doses of corticosteroids and at a stable dose of immunosuppressive drugs
* Indication for a seasonal influenza vaccination.

Existence of one or more of these clinical situations:

* pulmonary location (dyspnea, radiological or stage IV pulmonary function tests (PFT) altered with decreased forced vital capacity (FVC), forced expiratory volume average (FEV) or the diffusion of carbon monoxide (TLCO) below 65% of predicted value;
* Cardiac impairment confirmed
* Central nervous system impairment and / or device and confirmed with clinical impact and abnormal imaging and / or electromyogram- Renal impairment (histologically confirmed) responsible for a decrease in creatinine clearance
* disabling Lupus pernio
* Sinuso-nasal and / or laryngeal impairment histologically confirmed
* Disseminated impairment, ie affecting more than four organs
* Dose of corticosteroids ≥to 10 mg per day of the equivalent of prednisone or the necessity of an immunosuppressive therapy (with the exception of Rituximab) to control sarcoidosis- Existence of an associated metabolic disorder
* Patients with sarcoidosis and living in a care house
* Sarcoidosis occurring in health/nursing staff

Inclusion criteria for healthy volunteers

* Age ≥ 18 and ≤ 65 years
* Signature of informed consent
* Lack of underlying disease, especially autoimmune diseases and / or sarcoidosis
* Follow-up possible during the six months following the influenza vaccination

Exclusion Criteria for all:

* Hypersensitivity to the active substances, eggs and one of the excipients of the vaccine
* Acute febrile episode in the week prior to vaccination
* Count with a documented case of influenza within a week prior to vaccination
* Infection with HIV HBV or HCV known,
* Current pregnancy or positive urine pregnancy test
* Multiple Sclerosis
* History of Guillain-Barré
* Organ Transplantation
* Cancer in the last 3 years
* Other vaccination received within 3 weeks prior to the study vaccine injection
* Treatment with chemotherapy
* Transfusion or immunoglobulin administration during the last 3 months
* Co-morbidity requiring biological therapy that specifically targets B cells (eg rituximab)
* Patient for which an increase of the treatment is planned in the month following vaccination.
* Acute infection in the month prior to vaccination
* non affiliated to a health social security system
* Participation in another biomedical research for the duration of the study
* Individuals deprived of freedom by an administrative or court order

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Humoral immunogenicity | 21 days post-vaccination
  Humoral immunogenicity of the vaccine will be measured 3 weeks after injection of influenza vaccine (day 21) by comparison of the seroconversion rates between patients with sarcoidosis and the control group of healthy subjects.

SECONDARY OUTCOMES:
Immunogenicity | at Day 0, Day 21 and Day 180
  Effect of the initial clinical phenotype (including disease activity score) on the seroconversion and seroprotection rates, and the seroconversion factor, at each visit
Clinical phenotype | at Day 21 and Day 180
  Descriptive study of the evolution of clinical phenotype (eg, severity of illness) after vaccination at D21 and D180
Auto immunity activity | At Day 0, at Day 21 and at 6 months post-vaccination
  Comparison of autoantibody levels before and after vaccination (anti-nuclear total, rheumatoid factor, anti-GM1 measured at D0, D21 and D180) in all individuals included in the study.
Effect of therapy on immunogenicity | at Day 21 and Day 180
  Effect of the dose of corticosteroids and immunosuppressive therapy on the seroconversion and seroprotection rates and seroconversion factor at D21 and D180;
Immunogenicity between groups | at Day 0, Day 21 and Day 180
  Comparison of the seroprotection rate and the seroconversion factor between patients with sarcoidosis and the control group of healthy subjects at D21 and D180 post-vaccination.
Long term immune response | At 6 months post-vaccination
  Comparison of the persistence of the immune response between patients with sarcoidosis and control subjects at D180
Lymphocytes subpopulations analysis | At Day 0 and at 21 days post-vaccination
  Comparison between D0 and D21 of the distributions in absolute values and percentages of circulating lymphocyte subpopulations, in particular mucosal "homing" CD4+ lymphocytes, in all individuals included in the study;
Regulatory T Lymphocytes | At Day 0 and Day 21
  Effect of the regulatory T cells titers on the seroconversion and seroprotection rates, and the seroconversion factor at D0
Disease activity evolution | at Day 0, Day 21 and Day 180
  Effect of the CD4+-CD103+ T cells + at J0 and its evolution between J0 and J21 days based on the scalability of sarcoidosis evaluated by 1/changes in serum enzyme angiotensin converting, IgG, IgA IgM,; 2/ the comparative pulmonary radiological changes and 3/ the in pulmonary function changes between day 0 and day 180.
Other immune response | Between Day 0 to 6 months post-vaccination
  Seroprevalence and comparison between D0 and D180 of anti-diphtheria toxin and anti-tetanus toxin in all individuals included.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Le Jeunne, MD, PhD, Study Chair — Hôtel Dieu Hospital
Locations (1):
- Hotel-Dieu Hospital, Paris, France

REFERENCES:
- [Background] Mert A, Bilir M, Ozaras R, Tabak F, Karayel T, Senturk H. Results of hepatitis B vaccination in sarcoidosis. Respiration. 2000;67(5):543-5. doi: 10.1159/000067471. PMID 11070460
- [Background] Recommendation for the composition of influenza virus vaccines for use in 1999. Wkly Epidemiol Rec. 1998 Oct 2;73(40):305-8. No abstract available. English, French. PMID 9787645
- [Background] Statement on sarcoidosis. Joint Statement of the American Thoracic Society (ATS), the European Respiratory Society (ERS) and the World Association of Sarcoidosis and Other Granulomatous Disorders (WASOG) adopted by the ATS Board of Directors and by the ERS Executive Committee, February 1999. Am J Respir Crit Care Med. 1999 Aug;160(2):736-55. doi: 10.1164/ajrccm.160.2.ats4-99. No abstract available. PMID 10430755
- [Background] Bouvry D, Naccache JM, Valeyre D. [Interstitial lung diseases in sarcoidosis]. Rev Prat. 2007 Dec 31;57(20):2258-65. French. PMID 18320746
- [Background] Valeyre D, Duperron F. [Sarcoidosis: diagnosis and management of extra-pulmonary forms]. Rev Mal Respir. 2006 Dec;23(6):757-8. doi: 10.1016/s0761-8425(06)72092-7. No abstract available. French. PMID 17886354
- [Background] Lofgren S. The concept of erythema nodosum revised. Scand J Respir Dis. 1967;48(3):348-53. No abstract available. PMID 5183631
- [Background] James DG. Lupus pernio. Lupus. 1992 May;1(3):129-31. doi: 10.1177/096120339200100302. PMID 1301972
- [Background] Asukata Y, Ishihara M, Hasumi Y, Nakamura S, Hayashi K, Ohno S, Mizuki N. Guidelines for the diagnosis of ocular sarcoidosis. Ocul Immunol Inflamm. 2008 May-Jun;16(3):77-81. doi: 10.1080/09273940802051100. PMID 18569792